CLINICAL TRIAL: NCT05481008
Title: Cardiac Output, Cerebral Perfusion and Cognition in Patients With Severe Aortic Valve Stenosis Undergoing Transcatheter Aortic Valve Implantation
Brief Title: Cardiac Output, Cerebral Perfusion and Cognition in Patients Undergoing TAVI
Acronym: CAPITA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ronak Delewi (Other)
Responsible Party: Sponsor-Investigator, Ronak Delewi, MD PhD, Prinicipal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: NL72247.018.19
Record Dates: First submitted 2022-04-11; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Aortic Valve Stenosis; Cognitive Impairment; Cognitive Change
Keywords: Transcatheter aortic valve implantation; Aortic valve stenosis; Cognitive impairment; Cognition; Cerebral perfusion; Cerebral blood flow
MeSH Terms: conditions — Aortic Valve Stenosis; Cognitive Dysfunction | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: transcatheter aortic valve implantation — All subjects undergo transcatheter aortic valve implantation because of symptomatic severe aortic valve stenosis. This is a routine medical procedure, not a study intervention.

SUMMARY:
Rationale: Cardiovascular disease and cognitive diseases are closely related. Cognitive impairment is common (21-39%) among patients with severe aortic valve stenosis. The proof-of-concept CP-TAVI study showed that increased cardiac output following transcatheter aortic valve implantation (TAVI) was associated with increased cerebral blood flow. It is hypothesized that increased cerebral blood flow (CBF) subsequently leads to improved cognitive functioning. Additionally, silent micro emboli caused by crushing of the calcified native valve during TAVI may cause cognitive deterioration. If it could be predicted which patients are at risk for TAVI induced cerebral micro emboli, these patients could benefit from cerebral protection devices, preventing cognitive decline.

Objective: The objectives of the CAPITA study are 1A) to identify whether an increase in cardiac output after TAVI is associated with an increase of global CBF; 1B) explore regional differences in CBF after TAVI; 1C) determine whether (global or regional) increased CBF is associated with improved cognitive functioning; 1D) identify patient and procedural characteristics associated with increased cardiac output, CBF and cognitive functioning; 2A) identify the incidence and volume of new white matter hyperintensities after TAVI; 2B) evaluate patient and procedural predictors for the increase in white matter hyperintensities volume, including baseline aortic valve calcification volume, measured with computed tomography; 2C) if aortic valve calcification volume predicts new white matter hyperintensities, define a cut-off value for high-risk patients; 2D) assess whether the increase in white matter hyperintensity volume is associated with deterioration of cognitive scores.

Study design: Prospective observational study, measuring cardiac output (echocardiography), cerebral blood flow (arterial spin labelling magnetic resonance imaging) and cognitive functioning (neuropsychological test battery) prior to TAVI (<24 hours to <one week) and at 3 months follow-up. At one year follow-up, cardiac output and cognitive function will be assessed.

Study population: Patients with severe aortic valve stenosis eligible for transfemoral TAVI (n=142).

Main study parameters/endpoints: Cardiac output (L/min), cerebral blood flow (mL/100g/min, change in %, relative to baseline) and cognitive functioning (extensive neuropsychological testing 60-90 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic valve stenosis (aortic valve area <1cm2 and/or mean aortic valve gradient exceeds 50 mmHg) of a native valve
* Eligible for TAVI
* Able and willing to give informed consent
* Age > 18 years

Exclusion Criteria:

* Presence of MRI contra-indication; inability to lay flat for 30 minutes
* Weight > 130 kg
* Neurological disease
* Active malignant disease;
* Insufficient mastery of the Dutch language
* Inability to withdraw from alcohol use for 24 hours
* Non-atherosclerotic vascular disease (eg vasculitis)
* Planned surgery with general anesthesia within three months after TAVI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: N=142 patients with symptomatic severe aortic valve stenosis selected for transcatheter aortic valve implantation
Sampling Method: Non-Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Potential positive cerebral effects generated by an increase in cerebral blood flow after TAVI | Change from baseline (pre-tavi) to 3 months
  Cerebral blood flow (mL/100g/min, change in %, relative to baseline) as measured on arterial spin labelling magnetic resonance imaging)
Potential negative cerebral outcomes as a consequence of TAVI induced cerebral embolization | Change from baseline (pre-tavi) to 3 months
  New white matter hyperintensities (number and volume [mL]) and (micro) bleeds

SECONDARY OUTCOMES:
Cognitive functioning | Change from baseline (pre-tavi) to 3 months
  Cognitive functioning on various domains. As measured by a standardized extensive neuropsychological test battery (60-90 minutes) performed by a trained neuropsychologist.
Cognitive functioning | 1 year
  Cognitive functioning on various domains. As measured by a standardized extensive neuropsychological test battery (60-90 minutes) performed by a trained neuropsychologist.
Cardiac output | Change from baseline (pre-tavi) to 3 months
  Cardiac output (L/min) as measured on echocardiography (LVOT VTI)
Cardiac output | 1 year
  Cardiac output (L/min) as measured on echocardiography (LVOT VTI)

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam Universitair Medisch Centrum (AUMC) - Locatie AMC, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] van Nieuwkerk AC, Hemelrijk KI, Bron EE, Leeuwis AE, Majoie CBLM, Daemen MJAP, Moonen JEF, de Sitter A, Bouma BJ, van der Flier WM, Baan J, Piek JJ, Biessels GJ, Delewi R; Heart-Brain Connection Consortium. Cardiac output, cerebral blood flow and cognition in patients with severe aortic valve stenosis undergoing transcatheter aortic valve implantation: design and rationale of the CAPITA study. Neth Heart J. 2023 Dec;31(12):461-470. doi: 10.1007/s12471-023-01826-8. Epub 2023 Nov 1. PMID 37910335